CLINICAL TRIAL: NCT01690104
Title: The Effect of PXR Activation on Blood Pressure Regulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Rifa-BP; 2011-005522-22 (EudraCT Number)
Record Dates: First submitted 2012-09-07; First posted 2012-09-21 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2012-09

CONDITIONS: Blood Pressure Regulation
Keywords: rifampicin; pregnane X receptor; blood pressure
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifampicin (Active Comparator): Rifampicin 600 mg daily
  Interventions: Drug: Rifampicin
- Placebo (Placebo Comparator): Placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifampicin
  Other Names: Rimapen
  Arms: Rifampicin
Drug: Placebo
  Arms: Placebo

SUMMARY:
We are investigating the effects of pregnane X receptor (PXR) activation on the regulation of blood pressure in healthy volunteers. Rifampicin (an antibiotic and also an efficient PXR activator) and placebo will be given for a week to volunteers and blood pressure is measured 24 hours using an ambulatory blood pressure monitor. Blood pressure regulating hormones will be measured in blood. Our hypothesis is that PXR is involved in the regulation of blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BMI 19-30 kg/m2
* Age 18-40 years
* Systolic blood pressure 95 - 140 mmHg

Exclusion Criteria:

* Any continuous medication
* Any significant medical condition as judged by the study physician
* Diastolic blood pressure over 90 mmHg
* Sensitivity to rifampicin
* Pregnancy and lactation
* Difficult venipuncture
* Abuse of alcohol or medications, or drug use.
* Participation in other trial with medications in previous 30 days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Systolic ambulatory blood pressure | On day 8 of each arm
  Systolic blood pressure measured with ambulatory blood pressure monitor.
Diastolic ambulatory blood pressure | On day 8 of each arm
  Diastolic blood pressure measured with ambulatory blood pressure monitor

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | On day 9 of each arm
Pulse (ambulatory) | On day 8 of each arm
Plasma renin activity | On day 9 of each arm
Serum aldosterone | On day 9 of each arm

CONTACTS AND LOCATIONS:
Overall Officials: Janne Hukkanen, MD, PhD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Rahunen R, Kummu O, Koivukangas V, Hautajarvi H, Hakkola J, Rysa J, Hukkanen J. Pregnane X Receptor-4beta-Hydroxycholesterol Axis in the Regulation of Overweight- and Obesity-Induced Hypertension. J Am Heart Assoc. 2022 Mar 15;11(6):e023492. doi: 10.1161/JAHA.121.023492. Epub 2022 Mar 1. PMID 35229613